CLINICAL TRIAL: NCT01784419
Title: Short Term Effects of Ivacaftor in Non-G551D Cystic Fibrosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Screening
Other Study IDs: FS-001
Record Dates: First submitted 2013-02-03; First posted 2013-02-05 (Estimated); Results first posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Ivacaftor; Genotype; Phenotype; Sweat chloride; Pancreatic sufficient
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ivacaftor-placebo (Experimental): The ivacaftor-placebo arm receives a 2 week course of ivacaftor 150 mg twice daily followed by a 2 week washout period followed by a 2 week placebo course.
  Interventions: Drug: ivacaftor; Drug: Placebo
- placebo-ivacaftor (Experimental): The placebo-ivacaftor arm receives a 2 week placebo course followed by a 2 week washout period followed by a 2 week course of ivacaftor 150 mg twice daily.
  Interventions: Drug: ivacaftor; Drug: Placebo

INTERVENTIONS:
Drug: ivacaftor — Eligible subjects were randomized to ivacaftor 150 mg by mouth twice a day for 14 days followed by placebo for 14 days, or vice versa. Randomization was based on a computer-generated schedule produced by the research pharmacy, which was concealed from study personnel until study completion. Ivacaftor was purchased at full retail cost and encapsulated with sucrose to match the sucrose-filled placebo capsules. Prior to beginning study drug, there was a 2-week run-in period to ensure clinical stability, assessed by modified Fuchs criteria and pulmonary function. There was a washout period of a minimum of 14 days between study drug cycles to account for carryover effect. The washout period was extended to 6 weeks for subjects on alternating cycles of inhaled antibiotics to coordinate the study drug cycle with the inhaled antibiotic cycle.
  Other Names: Kalydeco; VX-770
Drug: Placebo — Eligible subjects were randomized to ivacaftor 150 mg by mouth twice a day for 14 days followed by placebo for 14 days, or vice versa. Randomization was based on a computer-generated schedule produced by the research pharmacy, which was concealed from study personnel until study completion. Ivacaftor was purchased at full retail cost and encapsulated with sucrose to match the sucrose-filled placebo capsules. Prior to beginning study drug, there was a 2-week run-in period to ensure clinical stability, assessed by modified Fuchs criteria and pulmonary function. There was a washout period of a minimum of 14 days between study drug cycles to account for carryover effect. The washout period was extended to 6 weeks for subjects on alternating cycles of inhaled antibiotics to coordinate the study drug cycle with the inhaled antibiotic cycle.

SUMMARY:
This is a study of the short-term effects of ivacaftor on sweat chloride concentration and lung function in cystic fibrosis (CF) patients who fall outside current FDA approval. This new, first of its kind drug is approved for use only in CF patients with the G551D mutation in whom it safely confers considerable benefits. However, it is highly likely that CF patients with many other mutations can benefit similarly from this drug, some of whom can be identified by phenotype or genotype.

We will enroll up to 30 CF subjects with clinical presentations in which there is one or more signs of residual CF channel function. The signs of residual function include: normal digestion, concentration of chloride in sweat between 55 and 85, or milder than expected CF disease in a CF patient with severe gene mutations. The primary outcome measure will be the difference in sweat chloride concentration measured in subjects on placebo and on ivacaftor. Secondary outcome measured will be lung function.

DETAILED DESCRIPTION:
Ivacaftor is a cystic fibrosis (CF)channel potentiator that is associated with decreased sweat chloride concentration, improved lung function, and improved weight gain. It is currently FDA approved for use only in CF patients with the G551D gating mutation. In vivo data suggest that ivacaftor may potentiate CF channels coded for by many other mutations associated with residual channel function, i.e., that some CF protein is present in the cell membrane of affected cells. This includes all of the 9 other known gating mutations, but ivacaftor also may be effective in CF patients with non-gating mutations, including some associated with severe phenotype. Based on results from previous studies, we hypothesize that non-G551D patients with signs of residual CF channel activity might respond favorably to treatment with ivacaftor. This includes patients with any of the non-G551D gating mutations, that are pancreatic sufficient, that have a sweat chloride concentration between 55 and 85 mmol, or that are much healthier than expected. Hence, select CF patients treated with ivacaftor as compared to placebo will have a decrease in sweat chloride concentration by greater than 20 mmol, improvement in FEV1, and weight gain. To test our hypothesis, we will conduct a prospective double-blinded placebo-controlled crossover clinical study comparing treatment with ivacaftor to placebo therapy (see details below). Our specific aims are:

Specific Aim 1: To demonstrate a decrease in sweat chloride concentration by greater than 20 mmol from baseline after 14 days of ivacaftor as compared to placebo.

Specific Aim 2: To demonstrate improvement in lung function measures from baseline after 14 days of Ivacaftor as compared to placebo.

Specific Aim 3:To demonstrate weight gain from baseline after 14 days of Ivacaftor as compared to placebo.

Study Design:

This is a prospective randomized double-blinded placebo-controlled crossover study of the short-term effects of ivacaftor (aka VX-770 or Kalydeco) on sweat chloride concentration and lung function in cystic fibrosis (CF) patients who fall outside current FDA approval.

We will enroll up to 30 CF subjects from the UCSF CF Center with a variety of genotypes and phenotypes in which there is one or more signs of residual CFTR function. The signs of residual CF channel function include: pancreatic sufficiency, sweat chloride concentration less than 85 mmol, or milder than expected CF disease in a CF patient with a severe genotype. We will exclude patients who are homozygous for the F508del mutation and have a sweat chloride concentration greater 85 mmol, which is true of the majority of F508del homozygotes. This population has been studied and found to be unresponsive to ivacaftor and includes nearly half of all CF patients. However, even among F508del homozygotes about 15 percent have residual chloride secretion manifest as a lower than expected sweat chloride concentration. The primary outcome measure will be the difference in sweat chloride concentration measured in subjects on placebo and on ivacaftor. Secondary outcome measures include variables obtained by spirometry and multi-breath washout testing.

Research Plan:

We will conduct a randomized double-blinded placebo-controlled crossover trial, in which all subjects will be treated with 2 weeks of ivacaftor and 2 weeks of placebo with a 2-week wash out period. Up to 30 subjects with one or more signs of residual CFTR function will be randomized into the study. This includes subjects who are pancreatic sufficient, who have a sweat chloride of 55 to 85 mmol, or who have mild CF disease in a setting of a severe CF genotype.

Each subject will act as his/her own control in a prospective randomized double-blinded crossover trial consisting of 14 days of ivacaftor or placebo, followed by a 14 day washout period, followed by 14 days of placebo or ivacaftor. The primary outcome measure will be sweat chloride concentration at baseline, 14 days, 28 days and 42 days. Secondary outcomes include standard lung function measures: forced vital capacity (FVC), forced expiratory volume at 1 second (FEV1), FEV1/FVC and mid-expiratory flow (FEF25-75), and multibreath washout testing. Blood samples will be examined at baseline, 14 days, 28 days and 42 days for evidence of drug toxicity (CBC with differential, liver function tests (AST, ALT), non-fasting glucose, creatinine and BUN). For female subjects of child bearing age, a urine pregnancy test will be done to assure they are not pregnant. If a female becomes pregnant during the study, the trial will be stopped but we will continue to measure sweat chloride, lung function, and blood work at the specified times. The effects of ivacaftor on the fetus are not known at this time.

Results of all laboratory tests will be forwarded to a nurse practitioner not directly involved with the study subjects, who will serve as the subject safety monitor. The nurse practitioner will notify study investigators of any laboratory values consistent with an adverse effect of study drug and will have the power to discontinue any subject in case of a serious adverse event. The most common serious adverse event in previous ivacaftor trials was mild elevation of liver tests. For this trial a serious adverse event sufficient to warrant discontinuing a subject will include a liver function test (ALT or AST) more than thrice the upper limit of normal, abnormal renal function or abnormal red or white cell counts.

ELIGIBILITY:
Inclusion Criteria:

* Two mutations known to cause cystic fibrosis and a sweat chloride concentration greater than or equal to 55 mmol
* Greater than or equal to 6 years of age

Exclusion Criteria:

* Homozygous F508del with a sweat chloride greater than 85 mmol
* Taking medication known to interact with ivacaftor and chooses not to discontinue that medication
* Is pregnant or planning to become pregnant during the study period
* Less than 6 years of age

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis W Nielson, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McGarry ME, Illek B, Ly NP, Zlock L, Olshansky S, Moreno C, Finkbeiner WE, Nielson DW. In vivo and in vitro ivacaftor response in cystic fibrosis patients with residual CFTR function: N-of-1 studies. Pediatr Pulmonol. 2017 Apr;52(4):472-479. doi: 10.1002/ppul.23659. Epub 2017 Jan 9. PMID 28068001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 72 patients were screened for eligibility.
Pre-assignment Details: All study participants are combined and reported here in one group because the data are reported this way in the only accessible data (in the publication). The PI has left the institution and the sequence specific data cannot be confirmed and are not available to be reported.
Groups:
- All Study Participants: The ivacaftor-placebo arm receives a 2 week course of ivacaftor 150 mg twice daily followed by a 2 week washout period followed by a 2 week placebo course.
  The placebo-ivacaftor arm receives a 2 week placebo course followed by a 2 week washout period followed by a 2 week course of ivacaftor 150 mg twice daily.
Period: Overall Study
Arm/Group | All Study Participants
Started | 10
Completed | 7
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5
  Persian | 1
  Latino | 1
Pancreatic sufficient [Count of Participants; unit: Participants] — Tests for pancreatic exocrine status, were used to determine pancreatic sufficiency or insufficiency status.
  Participants
    Yes | 5
    No | 2

OUTCOME MEASURES:

1. Primary Outcome: Sweat Chloride Concentration
Description: Sweat chloride concentration measured by pilocarpine iontophoresis, a standard clinical laboratory technique. Sweat collection accomplished with the Wescor Macroduct system. Sweat chloride is measured at the start and end of each study period. There are two study periods during which subjects take either ivacaftor or placebo.
Time Frame: 14 +/- 2 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
mmol/L | NA (NA) — The PI has left the institution and the only access to the data is from the publication. The access to this specific data cannot be confirmed and is not available to be reported.

2. Secondary Outcome: Spirometry
Description: Standard spirometry will be performed at the start and end of each 2 week study period. Subjects will take study drug (ivacaftor or placebo) during each study period.
Time Frame: 14 +/- 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Participants | NA — The PI has left the institution and the only access to the data is from publication. The access to this specific data cannot be confirmed and is not available to be reported.

3. Secondary Outcome: Multibreath Washout Testing
Description: Subjects will perform multibreath washout testing using standard techniques to measure functional residual capacity and lung clearance index at the beginning and end of each study period.
Time Frame: 14 +/- 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Participants | NA — The PI has left the institution and the only access to the data is from publication. The access to this specific data cannot be confirmed and is not available to be reported.

ADVERSE EVENTS:
Description: All study participants are combined and reported here in one group because the data are reported this way in the only accessible data (in the publication). The PI has left the institution and the sequence specific data cannot be confirmed and are not available to be reported.
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Study Participants (N=10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Injected conjunctiva (Eye disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Pulmonary exacerbations (Respiratory, thoracic and mediastinal disorders) | 2
Viral infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes